CLINICAL TRIAL: NCT06961188
Title: Clinical Study on Nanocrystalline Megestrol Acetate for Appetite Improvement and Weight Gain in First-Line Non-Squamous Non-Small Cell Lung Cancer Patients During Pre-Cachexia and Cachexia Stages.
Brief Title: Clinical Study on Nanocrystalline Megestrol Acetate for Appetite Improvement and Weight Gain in Pre-Cachexia and Cachexia Stages Key Terminology Analysis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Megaxia ES-NSCLC-01
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Metastatic (Stage IV) Non-squamous Non-small Cell Lung Cancer (Nsq-NSCLC) With Driver Gene Negativity; Untreated With Systemic Therapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanocrystalline Megestrol Acetate Oral Suspension (Experimental)
  Interventions: Drug: Nano-crystalline Megestrol Acetate Oral Suspension; Other: Standard Therapy
- No-Treatment Control (Active Comparator)
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Drug: Nano-crystalline Megestrol Acetate Oral Suspension — Nanocrystalline Megestrol Acetate Oral Suspension + Standard Therapy Nanocrystalline Megestrol Acetate Oral Suspension (125 mg/mL) was administered to the study group at 5 mL orally once daily (equivalent to 625 mg/day) until disease progression or completion of 12 weeks (maximum treatment duration: 12 weeks), whichever occurred first.
  Arms: Nanocrystalline Megestrol Acetate Oral Suspension
Other: Standard Therapy — Standard Therapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of nanocrystalline medroxyprogesterone acetate for improving appetite and weight gain patients with non-small cell lung cancer (NSCLC) and cachexia and pre-cachexia. The enrolled patients were those with advanced NSCLC who had not received therapy, negative for driver genes and ineligible for curative treatment, and were planned to receive PD-1 inhibitors in combination with platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years at the time of enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
* Life expectancy ≥6 months.
* Histologically or cytologically confirmed metastatic (stage IV) driver gene-negative non-squamous non-small cell lung cancer (NSCLC) that is unresectable and not amenable to curative therapy
* Subjects with no prior systemic chemotherapy for metastatic non-small cell lung cancer (NSCLC).

Exclusion Criteria:

* Presence of any gastrointestinal absorption-impairing conditions (e.g., dysphagia, malabsorption, prior gastrectomy, or uncontrolled vomiting); current use of tube feeding/parenteral nutrition; or existence of anorexia nervosa, psychiatric disorder-induced anorexia, or pain-related feeding intolerance.
* Driver gene-positive NSCLC or histologically/cytologically confirmed squamous cell-dominant NSCLC.
* Patients with Cushing's syndrome, adrenal/pituitary insufficiency; poorly controlled diabetes mellitus.
* Concurrent enrollment in another clinical trial, unless it is an observational/non-interventional study or the follow-up phase of an interventional trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of appetite improvement assessed by A/CS-12 (Anorexia/Cachexia Subscale of Functional Assessment of Anorexia/Cachexia Therapy) | Week 3
Proportion of individuals with weight gain exceeding 5% relative to baseline | Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China